CLINICAL TRIAL: NCT02241993
Title: The Accuracy Benefit of Dual vs Single Amperometric Glucose Sensors in Persons With Type 1 Diabetes: Effect of Inter-sensor Distance
Brief Title: The Multi-Sensor Distance Accuracy Study
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, W Kenneth Ward MD, Associate Professor, Oregon Health and Science University
Other Study IDs: 11619
Record Dates: First submitted 2013-11-06; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: glucose sensor; Inter-sensor distance
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 diabetic

SUMMARY:
The purpose of the study is to test the accuracy benefit of having two glucose sensors (over one sensor alone) when they are positioned: 2mm, 10mm, 20mm, or 30mm apart. It is not yet known how close two sensors can be and still work correctly.

DETAILED DESCRIPTION:
An artificial pancreas system will likely require multiple glucose sensing elements to function safely. It is not yet known how close two glucose sensors can be placed and still work properly. Meaning, if one is reading inaccurately,and the other is positioned adjacent to it, will it read inaccurately also, defeating the purpose of having two sensors. Twenty adult subjects with Type 1 diabetes will wear four Medtronic REAL-Time glucose sensors during two separate 10-hour studies. The inter-sensor distances of each pair to be tested will be: 2, 10, 20, and 30mm apart. The sensors will be inserted the day prior to the study day to allow for signal stabilization and calibration. During the study day, arterialized venous blood will be drawn every 15 minutes to measure blood glucose. The sensor values and interstitial values will be recorded from each sensor receiver at each time point. Subjects will be fed two standardized meals and given pre-meal insulin based on their typical insulin to carbohydrate ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes mellitus diagnosed for at least 6 months
2. Current usage of multiple daily injections or subcutaneous insulin pump treatment
3. Age 18-65 years
4. HbA1c of 6.0 - 9.5% at screening visit
5. BMI 21-35
6. Willingness to follow all study procedures, including attending all clinic visits
7. Willingness to sign informed consent and HIPAA documents

Exclusion Criteria: Subjects presenting with any of the following will not be included in the study.

1. Pregnancy or Lactation: for women of childbearing potential there is a requirement for a negative urine pregnancy test.
2. Renal insufficiency (serum creatinine of 2.0 mg/dL or greater). Serum ALT or AST equal to or greater than 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as a serum albumin of less the 3.3 g/dL; or serum bilirubin of over 2.
3. Hematocrit of less than or equal to 34%.
4. Congestive heart failure, NYHA class III or IV.
5. Visual impairment preventing reading of glucose meter values.
6. Active coronary artery disease as manifested by unstable angina, or a myocardial infarction or therapeutic coronary percutaneous procedure (e.g., PTCA, stent placement) or CABG within the past 4 months.
7. Active foot ulceration.
8. Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
9. Cerebrovascular accident within the past 6 months.
10. Active alcohol abuse, substance abuse, or severe mental illness (as judged by the principal investigator).
11. Active malignancy, except basal cell or squamous cell skin cancers.
12. Major surgical operation within 30 days prior to screening.
13. Seizure disorder (epilepsy).
14. Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
15. Currently administration of oral or parenteral corticosteroids.
16. Use of an investigational drug within 30 days prior to screening.
17. Bleeding disorder, treatment with warfarin, or platelet count below 50,000.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical practice Type 1 patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Difference between very large sensor accuracy errors (≥50% from reference glucose) with the simultaneous use of four sensors vs one sensor. | 9-hour collection period, X 2

SECONDARY OUTCOMES:
Difference between mean absolute relative difference with the simultaneous use of four sensors vs one sensor. | 9-hour glucose level collection, X 2

CONTACTS AND LOCATIONS:
Overall Officials: W. Kenneth Ward, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Ward WK, Casey HM, Quinn MJ, Federiuk IF, Wood MD. A fully implantable subcutaneous glucose sensor array: enhanced accuracy from multiple sensing units and a median-based algorithm. Diabetes Technol Ther. 2003;5(6):943-52. doi: 10.1089/152091503322640980. PMID 14709196
- [Background] Schmidtke DW, Pishko MV, Quinn CP, Heller A. Statistics for critical clinical decision making based on readings of pairs of implanted sensors. Anal Chem. 1996 Sep 1;68(17):2845-9. doi: 10.1021/ac9602027. PMID 8794921
- [Result] Castle JR, Engle JM, El Youssef J, Massoud RG, Yuen KC, Kagan R, Ward WK. Novel use of glucagon in a closed-loop system for prevention of hypoglycemia in type 1 diabetes. Diabetes Care. 2010 Jun;33(6):1282-7. doi: 10.2337/dc09-2254. Epub 2010 Mar 23. PMID 20332355